CLINICAL TRIAL: NCT02851693
Title: Study of Imaging Characteristics OCT of Skin Lesions Requiring Biopsy / Resection
Acronym: OCTSKIN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No open study.
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1608069; 2016-A00647-44 (Other: ANSM)
Record Dates: First submitted 2016-07-28; First posted 2016-08-02 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-03

CONDITIONS: Mixed Tumor, Malignant; Biopsy; Resection; Carcinoma; Keratosis
MeSH Terms: conditions — Mixed Tumor, Malignant; Carcinoma; Keratosis | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Optical Coherence Tomography (OCT) (Experimental)
  Interventions: Device: Optical Coherence Tomography (OCT) with Vivosight; Device: Optical Coherence Tomography (OCT) with Skintell

INTERVENTIONS:
Device: Optical Coherence Tomography (OCT) with Vivosight — OCT used is Vivosight for diagnosis
  Other Names: VIVOSIGHT (Michelson Diagnostics Ltd, Maidstone, Kent, UK)
Device: Optical Coherence Tomography (OCT) with Skintell — OCT used is Skintell for diagnosis
  Other Names: SKINTELL (Agfa HealthCare, Heverlee, Belgium)

SUMMARY:
The diagnosis of cutaneous lesions often involves the use of surgical and invasive procedures such as biopsy or excision in order to analyze the structure and appearance of the fabric pathologists. With recent advances in optical and electronic fields, considerable efforts were produced to build high-performance optical instruments, able to transcribe the internal structure of the skin with varying degrees of depth and variable resolution.

The imagery is now an area of great interest for medical diagnosis: non-invasive, quick, and in real time. This area is booming and new optical instruments are created to eventually be able to offer a reliable alternative to invasive techniques.

The optical properties of different tissues have been studied for several years by different research groups: the coefficient of light absorption by the tissue both in vivo and in vitro, the coefficient of light scattering or the index refractive were characterized in various tissues that make up the skin.

Other studies have focused on melanoma detection by multispectral optical techniques, or via the technique of optical coherence tomography (OCT) performed on lesions suspicious for cancer, but without linking criteria between these two techniques.

However, no study to date and to our knowledge has been able to demonstrate the different optical parameters obtained with OCT and can be directly connected to known and histopathological parameters commonly used in the diagnosis of lesions skin. This study aims to verify if it is possible to determine the parameters measured in OCT that would discriminate between benign and malignant lesions.

ELIGIBILITY:
Inclusion Criteria:

* patients with suspicious skin lesions of malignant tumor (mostly non-melanoma: basal cell carcinoma, epidermoid carcinoma and actinic keratoses, or melanoma: melanoma, nevi) requiring biopsy / surgical excision;
* consent signed

Exclusion Criteria:

* Any dermatosis, hyperalgesic lesion, and / or infected and / or topography making it impossible measurements;
* pregnant and nursing women
* patients under tutorship or curatorship

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
composite endpoint | at baseline
  thickness of the epidermis (µm), thickness of the dermis (µm), limit of epidermis/dermis, homogeneity of the epidermis, homogeneity and structure of the papillary dermis, vascular network associated, homogeneity of the reticular dermis, wall of vacuoles and nodules (presence or absence)

SECONDARY OUTCOMES:
implementation duration | at baseline
  minutes
acquisition practices duration | at baseline
  minutes
the duration of analysis image | at baseline
  minutes
utility of labeling with a dye for histology to locate the lesion | at baseline
  yes or no

CONTACTS AND LOCATIONS:
Overall Officials: Jean Luc PERROT, MD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne

IPD SHARING:
Plan to Share IPD: No